CLINICAL TRIAL: NCT02003807
Title: Incidence and Predictive Factor of Irritable Bowel Syndrome After Acute Diverticulitis in Korea
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0326
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Diverticulitis and Irritable Bowel Syndrome
MeSH Terms: conditions — Diverticulitis; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diverticulitis patients (case): Cases were the patients who admitted to hospital because of acute diverticulitis attack.
- Non-diverticulitis patients (control): Controls were the patients who admitted to hospital due to non-gastrointestinal disorder.

SUMMARY:
The pathogenesis of irritable bowel syndrome (IBS) is considered immune reaction of gastrointestinal tract. Therefore there is growing evidence that IBS could occur after gastroenteritis. However, little is known about the incidence of IBS after acute diverticulitis. We thought that post diverticulitis status could induce IBS because diverticulitis was also bowel inflammatory disorder. This survey was designed to identify incidence of post-diverticulitis IBS and risk factor in Korea.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or over
* Patients who diagnosed diverticulitis by CT scan from 2006 to 2010 (Case)
* Patients who admitted to hospital because of non-gastrointestinal disorder (Control)

Exclusion Criteria:

* Patients who diagnosed IBS before diverticulitis (Case)
* Patients who diagnosed IBS before admission (Control)
* Patients with bowel resection surgery except for laparoscopic appendectomy
* Pregnancy
* Do not agree the consent of this study
* Patients who dose not understand telephone survey such as foreigner, mental retardation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had admitted Severance hospital, Seoul, South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The newly developed IBS | Survey was done from 15th July 2013 to 30th September 2013
  The primary outcome was newly developed IBS. This was checked by telephone survey from 15th July 2013 to 30th September 2013. IBS was diagnosed by Rome III criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Ballou SK, Keefer L. Multicultural considerations in the diagnosis and management of irritable bowel syndrome: a selective summary. Eur J Gastroenterol Hepatol. 2013 Oct;25(10):1127-33. doi: 10.1097/MEG.0b013e3283632bf2. PMID 23778308
- [Background] Ohman L, Simren M. New insights into the pathogenesis and pathophysiology of irritable bowel syndrome. Dig Liver Dis. 2007 Mar;39(3):201-15. doi: 10.1016/j.dld.2006.10.014. Epub 2007 Jan 30. PMID 17267314
- [Background] Ishihara S, Tada Y, Fukuba N, Oka A, Kusunoki R, Mishima Y, Oshima N, Moriyama I, Yuki T, Kawashima K, Kinoshita Y. Pathogenesis of irritable bowel syndrome--review regarding associated infection and immune activation. Digestion. 2013;87(3):204-11. doi: 10.1159/000350054. Epub 2013 May 23. PMID 23712295
- [Background] Hughes PA, Zola H, Penttila IA, Blackshaw LA, Andrews JM, Krumbiegel D. Immune activation in irritable bowel syndrome: can neuroimmune interactions explain symptoms? Am J Gastroenterol. 2013 Jul;108(7):1066-74. doi: 10.1038/ajg.2013.120. Epub 2013 May 7. PMID 23649183
- [Background] Jung IS, Kim HS, Park H, Lee SI. The clinical course of postinfectious irritable bowel syndrome: a five-year follow-up study. J Clin Gastroenterol. 2009 Jul;43(6):534-40. doi: 10.1097/MCG.0b013e31818c87d7. PMID 19262407
- [Background] Zanini B, Ricci C, Bandera F, Caselani F, Magni A, Laronga AM, Lanzini A; San Felice del Benaco Study Investigators. Incidence of post-infectious irritable bowel syndrome and functional intestinal disorders following a water-borne viral gastroenteritis outbreak. Am J Gastroenterol. 2012 Jun;107(6):891-9. doi: 10.1038/ajg.2012.102. Epub 2012 Apr 24. PMID 22525306
- [Background] Ji S, Park H, Lee D, Song YK, Choi JP, Lee SI. Post-infectious irritable bowel syndrome in patients with Shigella infection. J Gastroenterol Hepatol. 2005 Mar;20(3):381-6. doi: 10.1111/j.1440-1746.2005.03574.x. PMID 15740480
- [Background] Spiller R, Garsed K. Postinfectious irritable bowel syndrome. Gastroenterology. 2009 May;136(6):1979-88. doi: 10.1053/j.gastro.2009.02.074. Epub 2009 May 7. PMID 19457422
- [Background] Strate LL, Modi R, Cohen E, Spiegel BM. Diverticular disease as a chronic illness: evolving epidemiologic and clinical insights. Am J Gastroenterol. 2012 Oct;107(10):1486-93. doi: 10.1038/ajg.2012.194. Epub 2012 Jul 10. PMID 22777341
- [Background] Cohen E, Fuller G, Bolus R, Modi R, Vu M, Shahedi K, Shah R, Atia M, Kurzbard N, Sheen V, Agarwal N, Kaneshiro M, Yen L, Hodgkins P, Erder MH, Spiegel B. Increased risk for irritable bowel syndrome after acute diverticulitis. Clin Gastroenterol Hepatol. 2013 Dec;11(12):1614-9. doi: 10.1016/j.cgh.2013.03.007. Epub 2013 Mar 21. PMID 23524129
- [Background] Rafferty J, Shellito P, Hyman NH, Buie WD; Standards Committee of American Society of Colon and Rectal Surgeons. Practice parameters for sigmoid diverticulitis. Dis Colon Rectum. 2006 Jul;49(7):939-44. doi: 10.1007/s10350-006-0578-2. No abstract available. PMID 16741596
- [Background] Hammond NA, Nikolaidis P, Miller FH. Left lower-quadrant pain: guidelines from the American College of Radiology appropriateness criteria. Am Fam Physician. 2010 Oct 1;82(7):766-70. PMID 20879699
- [Background] Thabane M, Kottachchi DT, Marshall JK. Systematic review and meta-analysis: The incidence and prognosis of post-infectious irritable bowel syndrome. Aliment Pharmacol Ther. 2007 Aug 15;26(4):535-44. doi: 10.1111/j.1365-2036.2007.03399.x. PMID 17661757
- [Background] Spiller R. Is it diverticular disease or is it irritable bowel syndrome? Dig Dis. 2012;30(1):64-9. doi: 10.1159/000335721. Epub 2012 May 3. PMID 22572688
- See also: Official web site of Rome Foundation. The definition of IBS and questionnaire was adopted from that web site. — http://www.romecriteria.org/